CLINICAL TRIAL: NCT06171815
Title: University of Health Sciences, Hamidiye Faculty of Nursing
Brief Title: Comparison of Peer-Led Simulation Facilitation Methods on Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Associate Proffessor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023/16-25
Record Dates: First submitted 2023-11-21; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Simulation of Physical Illness; Nurse's Role
Keywords: simulation, peer-led, facilitation

STUDY DESIGN:
Intervention Model Description: This research is a prospective, randomized, crossover-designed experimental type research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Arm (Experimental): Students in the first arm received simulation training under the leadership of a peer facilitator on the first day, and under the leadership of an instructor facilitator on the second day.
  Interventions: Behavioral: Scenario-based simulation
- Second Arm (Experimental): Students in the second arm received simulation training under the leadership of an instructor facilitator on the first day and under the leadership of a peer facilitator on the second day.
  Interventions: Behavioral: Scenario-based simulation

INTERVENTIONS:
Behavioral: Scenario-based simulation — Scenario-based simulation prepared for Respiratory Activity and Diabetes Management topics in the course curriculum

SUMMARY:
There are limited studies in the literature on the peer-led facilitator involved in each stage of the simulation in simulation-based experience in nursing education. The purpose of this research is to examine the effect of having a competent senior nursing undergraduate student with simulation knowledge and experience as a facilitator at every stage of the simulation, on the effectiveness of the simulation (Simulation Effectiveness Tool), and on the participants' satisfaction and self-confidence in learning.

Method: This research is a prospective, randomized, crossover-designed experimental type of research. Structured Student Information Form, Modified Simulation Effectiveness Tool, Student Satisfaction, and Self-Confidence in Learning Scale will be used to collect data. The population of the research consists of all students enrolled in the first year of the Hamidiye Faculty of Nursing at the University of Health Sciences. Since voluntary participation in the research is based, students who want to participate will constitute the sample. Students will be divided into two groups of eight and will undergo two simulations for two consecutive days. Students in the first arm completed the simulation under the leadership of a peer facilitator on the first day, and under the leadership of an instructor facilitator on the second day; Students in the second arm will receive simulation training under the leadership of an instructor facilitator on the first day, and under the leadership of a peer facilitator on the second day.

DETAILED DESCRIPTION:
The instructor who facilitates the simulation training has a "Simulation Applications" certificate. The peer facilitator is a 4th-grade student who has received 2-day simulation training and has at least 3 simulation experiences.

Students will be divided into two groups of eight and will undergo two simulations for two consecutive days. Students in the first arm completed the simulation under the leadership of a peer facilitator on the first day, and under the leadership of an instructor facilitator on the second day; Students in the second arm will receive simulation training under the leadership of an instructor facilitator on the first day, and under the leadership of a peer facilitator on the second day.

In this study, data will be collected through a 3-stage application process.

1. Information

   * Respiratory Activity and Diabetes Management topics, which are in the Health Assessment course curriculum, will be explained to first-year students in the spring semester of the 2023-2024 Academic Year at the Faculty of Nursing, where the study will be carried out, by the instructor in charge of the course on the days and hours specified in the course program.
   * At the end of the course, explain to the students the purpose of the study, the method, and that the data will be used only for scientific purposes.
   * Students who volunteer to participate in the study are explained to the students who volunteer to participate in the study, and their verbal and written consent is obtained by explaining the duration, flow, and expectations of the application.
   * Informing students by deciding on the application day and time
   * Providing orientation to students by giving them information about the simulation environment and management in the application laboratory on the application day.
2. Simulation Training

   * Sharing the patient's information for which a scenario text was created for the students before the application.
   * Explaining what the goals are expected from students.
   * Carrying out both simulation applications on separate days and in a way that students in both groups stay in the simulation environment for the same amount of time.
3. Analysis

   * Holding a peer evaluation meeting after the simulation, where the groups experience the simulation.
   * Discuss students' thoughts about the process (their practices, decisions, and outcomes) regarding their simulation experience.
   * Discussing expected and achieved goals.
   * Following the analysis meeting, the Structured Student Information and Evaluation Form, Modified Simulation Effectiveness Tool, Student Satisfaction, and Self-Confidence in Learning Scale are administered to the students.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Having taken the Health Assessment course,
* Experienced education with simulation for the first time,
* Being willing and able to participate in the study.

Exclusion Criteria:

* Incomplete filling of Data Collection Forms,
* Not attending the simulation training on the day and time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Simulation Effectiveness | Through study completion, an average of 1 months
  Output regarding students' perceptions of the effectiveness of learning in a simulation environment. It will be measured with the Modified Simulation Effectiveness Tool. The measurement tool has 19 items and four subscales. Sub-dimensions of the measuring tool; These are prebriefing, learning, confidence and debriefing. The preliminary information sub-dimension consists of two items, the learning sub-dimension consists of six items, the trust sub-dimension consists of six items, and the analysis sub-dimension consists of five items.
Student Satisfaction and Self-Confidence in Learning | Through study completion, an average of 1 months
  Outcome regarding students' attitudes and beliefs about simulation. It will be measured by the Student Satisfaction and Learning Self-Confidence Scale. The scale, which is widely used to measure students' attitudes and beliefs about simulation, was published by the National League for Nurses (NLN) (Franklin, Burns and Lee 2014). It consists of two subscales: "satisfaction with learning" and "self-confidence" and a total of 13 items. In the satisfaction with learning sub-dimension; Five items measuring satisfaction with the teaching method, variety of learning materials, facilitation, motivation and overall suitability of the simulation are included in the self-confidence subscale; There are eight sub-items in content adequacy: self-confidence, content necessity, skill development, available resources and information on how to get help to solve clinical problems in the simulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Niu Y, Liu T, Li K, Sun M, Sun Y, Wang X, Yang X. Effectiveness of simulation debriefing methods in nursing education: A systematic review and meta-analysis. Nurse Educ Today. 2021 Dec;107:105113. doi: 10.1016/j.nedt.2021.105113. Epub 2021 Aug 27. PMID 34492539